CLINICAL TRIAL: NCT04710485
Title: Spheno_orbital Meningioma Enplaque With Proptosis; Surgical Techniques and Outcomes
Brief Title: Sphenoorbital Meningioma Management.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa metwally kashef ali, Assistant lecturer, Assiut University
Other Study IDs: Mng
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Brain Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators will discuss the different surgical techniques for removal of spheno_orbital meningiomas with proptosis.investigators also will follow up the patient to know the outcome of removal of these tumours.

ELIGIBILITY:
Inclusion Criteria:

* all patients who have spheno_orbital meningioma with proptosis and candidate for surgery.

Exclusion Criteria:

* all patients have proptosis caused by other lesions than spheno_orbital meningioma.

Ages: 5 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Any patient candidate for surgery will be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-01-30 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment for vision. | For 6 months
  With visual acuity examination
Clinical assessment for proptosis | For 6 months
  With proptosis index

CONTACTS AND LOCATIONS:
Overall Officials: Assiut Au University, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided